CLINICAL TRIAL: NCT01822977
Title: The Impact of Proton Pump Inhibitors on the Fecal Microbiome and Their Relationship to Clostridium Difficile Infection
Brief Title: The Impact of Proton Pump Inhibitors on the Fecal Microbiome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, John K. DiBaise, PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 13-000180
Record Dates: First submitted 2013-03-26; First posted 2013-04-04 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Healthy; Clostridium Difficile Infection
Keywords: gut microbiota; proton pump inhibitor; Clostridium difficile infection; Fecal microbiome; single episode of CDI
MeSH Terms: conditions — Clostridium Infections | interventions — Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Proton pump inhibitor (No Intervention): We will recruit 10 healthy adult individuals and 5 adult patients with an initial episode of CDI cared for at Mayo Clinic in Arizona. A baseline stool sample will be collected from the healthy individuals. They will then be given a PPI, omeprazole 20 mg, to be taken once (n=5) or twice (n=5) daily for 1 month. Stool samples will be collected after 1 week and again after 1 month. A final stool sample will be collected 1 month after stopping the omeprazole.
  A stool sample will be collected from the CDI subjects before treatment of the infection and again 2 months after treatment to avoid enrolling those at risk for relapse (which most commonly occurs during the first 2 months after treatment).
  Interventions: Drug: omeprazole

INTERVENTIONS:
Drug: omeprazole

SUMMARY:
The investigators hypothesis is that daily use of a proton pump inhibitor (PPI) is associated with significant alterations in the healthy fecal microbiome that are similar to those seen in persons with an initial episode of clostridium difficile infection (CDI).

ELIGIBILITY:
Table 1. Inclusion Criteria for Healthy Volunteers:

1. Healthy individuals without chronic gastrointestinal problems or using antisecretory medications.

Table 2. Inclusion Criteria for Clostridium difficile infection subjects:

1. Newly diagnosed first episode of CDI prior to being treated.

Table 3. Exclusion Criteria for Healthy Subjects:

1. Prior gastrointestinal surgery that has altered the anatomy of the esophagus, stomach, or small/large intestine including appendectomy and cholecystectomy.
2. Chronic daily use of any medications that could alter gastrointestinal secretory or motor function (see Table 2).
3. Gastrointestinal, cardiovascular, endocrine, renal, or other chronic disease likely to affect gastrointestinal motility (e.g., uncontrolled diabetes mellitus).
4. Females of childbearing age who are not practicing at least one form of birth control at least one month prior to starting the PPI or are pregnant or lactating (a pregnancy test will be performed on female subjects prior to PPI use).
5. Significant untreated psychiatric disease.

Table 4. Prohibited Medications:

1. Antibiotics within 2 months of the stool sample collection.
2. Probiotics (e.g., Florastor, Align, Flora-Q, VSL#3, lactobacillus, bifidobacterium) within 2 weeks of the stool sample collection.
3. Fiber supplements (e.g., Metamucil, Citrucel, Benefiber), unless maintained on a stable dose for the last 3 months.
4. Chronic use of medications that alter gastric pH: proton pump inhibitors (e.g., omeprazole, lansoprazole, esomeprazole, pantoprazole, rabeprazole, dexlansoprazole) and histamine2 receptor antagonists (e.g., cimetidine, famotidine, ranitidine).
5. Chronic use of medications that affect gastrointestinal motility and/or transit including prokinetic agents (e.g., metoclopramide (Reglan), tegaserod (Zelnorm), domperidone (Motilium), erythromycin), narcotic analgesic agents (e.g., methadone, fentanyl, oxycodone, codeine, morphine, hydromorphone), laxatives including mineral oil, anticholinergic agents (e.g., Bentyl, Levsin), and antidiarrheal agents (e.g., Kaopectate (donnagel), Pepto-Bismol (bismuth subsalicylate), Imodium (loperamide), Lomotil (atropine with diphenoxylate), codeine, tincture of opium).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Changes in fecal microbial diversity due to PPI therapy | 2 months

SECONDARY OUTCOMES:
Changes in fecal microbial diversity due to CDI | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: John Di Baise, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States